CLINICAL TRIAL: NCT00002232
Title: GENEVAX-HIV (APL 400-003), a Candidate DNA Vaccine: A Pilot Study of GENEVAX-HIV Given by Intramuscular or Intradermal Administration in HIV Seronegative Volunteers
Brief Title: A Study of GENEVAX-HIV, a Possible Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth-Lederle Vaccines (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Prevention
Other Study IDs: 005; 400-003-05
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Injections, Intradermal; Injections, Intramuscular; HIV Antibodies; Immunity, Cellular; AIDS Vaccines; HIV Seronegativity; Dose-Response Relationship, Immunologic; Vaccines, DNA; Immunity, Mucosal
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: APL 400-003

SUMMARY:
The purpose of this study is to see if it is safe to give GENEVAX-HIV, a potential HIV vaccine, to HIV-negative volunteers. The study also compares the effects of GENEVAX-HIV injected into the muscle to the effects of the drug when injected into the skin.

DETAILED DESCRIPTION:
Volunteers receive either intradermal or intramuscular injections of GENEVAX-HIV; humoral and cellular responses are assessed accordingly.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Good health.
* Ability to understand the basis of HIV transmission and other common sexual and blood-borne infections.
* The following parameters within normal range:
* Hematopoietic:
* total white blood cell, lymphocyte, granulocyte, and platelet count, hemoglobin and hematocrit.
* Renal:
* BUN and creatinine, urinalysis.
* Hepatic:
* total serum bilirubin.
* Endocrine/Metabolic:
* Serum calcium, serum glucose, total serum CPK.
* Immunologic:
* total serum immunoglobulin and absolute CD4 count.
* Hepatitis B and Hepatitis C negative.
* Urinalysis:
* Normal screen with dipstick for esterase and nitrite.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* HIV-seropositive status.
* Any positive result for anti-DNA antibodies considered of potential clinical significance as measured by anti-DNA antibody and/or anti-nuclear antibody (ANA) assays.
* Any condition which, in the opinion of the principal investigator, might interfere with completion of the study or evaluation of the results.
* Known hypersensitivity to bupivacaine or any amide-type local anesthetic (such as lidocaine, dibucaine, mepivacaine, and prilocaine) or a history of anaphylaxis or other serious adverse reactions to vaccines.

Concurrent Medication:

Excluded:

Any medication which may affect immune function with the exception of low doses of nonprescription-strength NSAIDS, aspirin, or acetaminophen for acute conditions such as headache or trauma.

Patients with the following prior conditions are excluded:

* HIV-seropositive.
* Known or suspected history of impairment or abnormality in immune functioning.
* Exposure to potentially-infective HIV fluids within the prior 6 months or tested positive for HIV at any time.
* History of any prior disease or therapy which would affect immune function including:
* Prior malignancy, except curatively-treated basal cell or squamous cell carcinoma in situ of the cervix.
* Immunodeficiency or autoimmune disease.
* Acute infection or a recent (within 6 months) history of chronic infection.
* History of serious allergic reaction to any substance requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).

Prior Medication:

Excluded:

Cytotoxic chemotherapy that may affect immune function.

Prior Treatment:

Excluded:

* Previous immunization with any experimental vaccines directed against HIV or receipt of any experimental agent within 30 days prior to enrollment.
* Receipt of any blood products or immunoglobulin within 6 months prior to enrollment.
* Exposure to live attenuated vaccines within 60 days of study.
* Radiotherapy that may affect immune function.

Risk Behavior:

Excluded:

* Active drug or alcohol abuse or uncontrolled (unstable) psychiatric disorders which, in the opinion of the investigator, would interfere with study participation.
* Higher- or intermediate-risk sexual behavior (AVEG criteria)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Merlin Robb, Study Chair
Locations (1):
- Walter Reed Army Institute of Research, Washington D.C., District of Columbia, United States